CLINICAL TRIAL: NCT02753244
Title: A Study to Assess the Feasibility of Intendu Cognitive Motion-Based Videogames in Acquired Brain Injury Patients and to Evaluate the Effects of Training on Their Cognitive Performance
Brief Title: Cognitive Motion-Based Videogames Exploratory Study in Acquired Brain Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Intendu Ltd. (Industry)
Collaborators: Tel Aviv University (Other); Sheba Medical Center (Other Government); Loewenstein Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00070-001; 2215 - 15 - SMC (Other: Sheba Medical Center)
Record Dates: First submitted 2016-04-10; First posted 2016-04-27 (Estimated); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Acquired Brain Injury
Keywords: Cognitive VideoGames
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Intendu FBT inpatient (Experimental): Other: Motion Based Cognitive Video Games Software
  Interventions: Other: Motion Based Cognitive Video Games Software
- iPad games (Active Comparator): Other: iPad apps
  Interventions: Other: iPad Apps
- Intendu FBT community (Experimental): Other: Motion Based Cognitive Video Games Software
  Interventions: Other: Motion Based Cognitive Video Games Software

INTERVENTIONS:
Other: Motion Based Cognitive Video Games Software — Intendu FBT motion based cognitive video games software
  Arms: Intendu FBT community; Intendu FBT inpatient
Other: iPad Apps — Commercially available iPad game applications
  Arms: iPad games

SUMMARY:
This study aims to assess the feasibility of Intendu Cognitive Motion-Based Videogames in Acquired Brain Injury (ABI) patients in inpatient treatment and in the community and to evaluate the effects of training on patients' cognitive performance

DETAILED DESCRIPTION:
This study includes three experimental arms to research cognitive video games involving motion interaction in ABI population. The study consists of 4 primary phases: recruitment, assessment, intervention and post-intervention assessment. Two arms involve a randomized controlled study with inpatient participants, where participants are randomly assigned to an intervention or control group. Recruitment phase includes cognitive assessments to evaluate eligibility for the study. In the assessment and post assessment phases cognitive performance is established.

Intervention includes 10 computerized training sessions of 30-45 minutes over 3 weeks period using Intendu Functional Brain Trainer (FBT). The control group intervention involves playing commercial iPad games for the same duration. Interventions will be performed in addition to standard inpatient treatment.

In addition to the randomized control study, a third experimental arm will be performed, were participants living in the community will perform a similar protocol with cognitive motion-based video games. The recruitment, assessment, post assessment and intervention phases will be similar to the above.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with Acquired Brain Injury.
2. At least one functional upper limb.
3. Ability to understand instructions that will be assessed by the therapist.
4. Basic cognitive ability in Orientation, Visual Perception and Spatial Perception.
5. Impairment in Executive Functions (EF) as assessed by EF assessments.
6. normal vision.

Exclusion Criteria:

1. Untreated epilepsy
2. Other Psychiatric or Neurological disease.
3. Neglect or Hemianopia.
4. For the Community arm - doesn't receive any cognitive therapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-04; Primary Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Change in Cognitive Functions | Week 0, week 4
  Assessments of cognitive skills as they express in task performance.
Change in Cognitive Performance Questionnaires | Week 0, week 4
  Questionnaire assessing cognitive skills as they express in everyday function.

SECONDARY OUTCOMES:
Experience during intervention | week 4
  Questionnaire regarding experience from intervention (e.g. satisfaction, exertion, etc.) following training.
Safety - Record of any adverse event | Weeks 0-4
  Any adverse event occurring during or following the intervention will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Ofer Keren, MD, Principal Investigator — Sheba Medical Center; Yaron Sacher, MD, Principal Investigator — Loewenstein Hospital
Locations (2):
- Israel (2):
  - Traumatic Brain Injury department, Loewenstein Hospital, Raanana
  - The Sheba Rehabilitation Hospital, The Head Trauma Rehabilitation Department, Ramat Gan

IPD SHARING:
Plan to Share IPD: No